CLINICAL TRIAL: NCT01865786
Title: A Prospective, Observational Study of Pregnancy Outcomes Among Women Exposed to Truvada for PrEP Indication Nested in the Antiretroviral Pregnancy Registry
Brief Title: A Prospective, Observational Study of Pregnancy Outcomes Among Women Exposed to Truvada for PrEP Indication
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-276-0101
Record Dates: First submitted 2013-05-22; First posted 2013-05-31 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: HIV Infection
Keywords: FTC/TDF; Truvada; PrEP; Antiretroviral Pregnancy Registry
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FTC/TDF for PrEP: The study has one target prospective cohort defined as HIV-1 negative women who had been prescribed FTC/TDF for pre-exposure prophylaxis (PrEP); with two strata: a) those who continue to take FTC/TDF for PrEP during their pregnancy, and b) those who decide to stop FTC/TDF for PrEP during pregnancy.
- ARV population: The study has one comparison cohort defined as HIV-positive women who were on any antiretroviral (ARV) medication at the time the pregnancy was detected. This is a propensity score matched retrospective cohort selected from the prospective arm of the APR. This cohort is assembled retrospectively in order to appropriately match the subjects by calendar time and the correlates of exposure, with exposure being defined as being on FTC/TDF for PrEP vs being exposed to other ARVs.

SUMMARY:
This is a prospective, observational study to describe pregnancy outcomes among HIV-1 uninfected pregnant women who are taking emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF) (Truvada®) for a pre-exposure prophylaxis (PrEP) indication nested in the Antiretroviral Pregnancy Registry (APR).

Information on subjects is provided to the APR prospectively (prior to the outcome of the pregnancy being known) through their healthcare provider, with follow-up obtained from the healthcare provider following determination of the pregnancy outcome.

ELIGIBILITY:
Key Inclusion Criteria:

* Pregnant women
* Part of the prospective arm of the APR Target Group Inclusion Criteria
* HIV-1 Negative
* Choosing to remain on FTC/TDF for PrEP during pregnancy or,
* Choosing to discontinue FTC/TDF for PrEP during pregnancy Comparison Group Inclusion Criteria
* HIV-1 Positive
* On antiretroviral therapy

Key Exclusion Criteria:

* This is an observational nested study and will monitor all reported exposures without intervention/exclusion.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Number of Subjects and Subject Selection: 400 HIV-1 uninfected women who are exposed to FTC/TDF for PrEP during pregnancy stratified into 200 who decide to continue and 200 who choose to discontinue FTC/TDF for PrEP. A propensity score-matched comparison group of equal size (400 women) of HIV-positive pregnant women taking antiretrovirals.
  All evaluable subjects enrolled into the APR who fulfill the inclusion criteria for the target cohort will be selected. Every year at the time of building the annual report for this study, a propensity score matched comparison group will be selected on a 1:1 ratio among all pregnant women on antiretrovirals.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-13 (Actual)

PRIMARY OUTCOMES:
Presence or absence of congenital malformations among infants born to HIV-1 uninfected women on FTC/TDF for PrEP | Year 1

SECONDARY OUTCOMES:
Pregnancy outcomes in HIV-1 uninfected women who choose to continue or discontinue FTC/TDF for PrEP during their pregnancy as well as HIV-infected women treated with antiretrovirals | Years 1, 2, and 3

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (1):
- Antiretroviral Pregnancy Registry, Wilmington, North Carolina, United States